CLINICAL TRIAL: NCT01135849
Title: B-Receptor Signaling in Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: Daniel Bernstein (Other)
Responsible Party: Sponsor-Investigator, Daniel Bernstein, Professor, Stanford University
Organization: Stanford University (Other)
Other Study IDs: PEDSVAR0038; SU-11172008-1345 (Other: Stanford University)
Record Dates: First submitted 2010-06-01; First posted 2010-06-03 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Carcinomas; Amyloidosis; Anal Cancer; Anemia; Cholangiocarcinoma of the Extrahepatic Bile Duct; Transitional Cell Carcinoma of Bladder; Bone Marrow Transplant Failure; Bone Cancer; Cancer of Brain and Nervous System; Breast Cancer; Carcinoma of the Large Intestine; Endocrine Cancer; Esophageal Cancer; Eye Cancer; Gall Bladder Cancer; Gastric (Stomach) Cancer; Gastrooesophageal Cancer; Gastrointestinal Stromal Tumor (GIST); Gynecologic Cancers; Head and Neck Cancers; Hepatobiliary Neoplasm; Kidney (Renal Cell) Cancer; Leukemia; Lung Cancer; Hodgkin Disease; Lymphoma, Non-Hodgkin; Mesothelioma; Multiple Myeloma; Myelodysplastic Syndromes (MDS); Neuroendocrine Tumors; Myeloproliferative Disorders; Pancreatic Cancer; Prostate Cancer; Skin Cancer; Soft Tissue Sarcoma; Testicular Cancer; Thymus Cancer; Thyroid Cancer
MeSH Terms: conditions — Carcinoma; Amyloidosis; Anus Neoplasms; Anemia; Bone Neoplasms; Brain Neoplasms; Neurologic Manifestations; Breast Neoplasms; Colonic Neoplasms; Endocrine Gland Neoplasms; Esophageal Neoplasms; Eye Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Gastrointestinal Stromal Tumors; Head and Neck Neoplasms; Carcinoma, Renal Cell; Leukemia; Lung Neoplasms; Hodgkin Disease; Lymphoma, Non-Hodgkin; Mesothelioma; Multiple Myeloma; Myelodysplastic Syndromes; Neuroendocrine Tumors; Myeloproliferative Disorders; Pancreatic Neoplasms; Prostatic Neoplasms; Skin Neoplasms; Sarcoma; Testicular Neoplasms; Thymus Neoplasms; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — cheek swab or blood drawn for DNA extraction
Oversight: Data Monitoring Committee: Yes

SUMMARY:
We hope to determine the importance of different genes (including B receptors) in anthracycline-induced cardiomyopathy. This has important benefits to patients exposed to anthracyclines, as this could help determine whether certain individuals have increased susceptibility to cardiac injury.

DETAILED DESCRIPTION:
There is a strong correlation between total doxorubicin dose and anti-tumor efficacy, however, the clinical utility of doxorubicin is severely limited by its cardiotoxicity. With improved methods of detecting subtle changes in cardiac function, e.g. alterations in left ventricular wall stress (1), the incidence of doxorubicin cardiotoxicity is now appreciated to be much higher than previously suspected, documented in 65% of long-term survivors of childhood cancer, even at doses as low as 228 mg/m2. This cardiotoxicity is dose-related, and higher doses are related to a higher incidence of clinical heart failure (2). Doxorubicin's cardiotoxicity is thought to be mediated through the generation of free radicals and through mitochondrial and membrane damage.

We wish to determine whether beta-receptor genotype affects anthracycline-induced cardiomyopathy. We will correlate beta-receptor genotype with difference in wall stress post-anthracycline exposure, and with difference in shortening fraction. We plan to recruit 300 patients over a two-year period. Inclusion criteria includes past exposure to anthracycline for cancer treatment and an echocardiogram 6 - 48 months after exposure to anthracyclines.

The mean difference in 1.) wall stress and 2.) shortening fraction between each minor allele subgroup and wild type subgroup, for both beta-1 and beta-2 will be assessed using unpaired t-test analyses . We will assess through multivariate linear regression whether there are interactions between differences in wall stress or fractional shortening and other variables such as age, gender, dose of anthracycline, type of anthracycline given, and time between anthracycline exposure and echocardiogram. Those who receive other cardiotoxic drugs (such as trastuzumab for breast cancer) will be analyzed separately.

ELIGIBILITY:
Inclusion Criteria:1.) Past exposure to anthracycline chemotherapy for cancer

2.) Echocardiogram at least six months after exposure to anthracyclines (in patients over the age of 40, the echocardiogram must be obtained within 6 - 48 months of anthracycline exposure)

3.) Ability to understand and the willingness to sign a written informed consent document.

We have no age, gender, or ethnic background limitations. Due to the increased frequency of cardiovascular disease from other causes in adults over 40 years, we will limit enrollment to those patients with an echocardiogram 6 - 48 months after the completion of anthracycline exposure. Children will be included and will be eligible if they have an echocardiogram at least 6 months after completion of anthracycline treatment..

Exclusion Criteria:1.) Congenital heart disease (other than patent foramen ovale)

2.) Pre-existing cardiomyopathy before anthracycline administration

3.) Patients with Down syndrome

4.) Patients receiving B-blocker therapy at the time of anthracycline exposure

5.) Pregnant patients (if their echocardiogram was obtained either during pregnancy or within three months of pregnancy)

All participants will be cancer survivors. To minimize bias from post-partum cardiomyopathy, pregnant patients will be excluded if their echocardiogram was obtained during pregnancy or within three months of pregnancy. HIV-positive persons will not be excluded from the study.

Of note, some patients receive a MUGA (multigated acquisition) study to evaluate left ventricular ejection fraction. Patients who receive only a MUGA scan will NOT be included in the study - an echocardiogram is necessary

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients exposed to anthracycline who have had an echocardiogram at least six months after initial exposure.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Development of cardiomyopathy | Within 5 years after receiving anthracyclines.
  Decrease in fractional shortening below normal (<28%)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bernstein, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States